CLINICAL TRIAL: NCT02239419
Title: Evaluation of the Clinical Utility, Efficacy and Safety of a Novel Medical Device (Carbothera) in the Treatment of Foot Ulcers
Brief Title: Evaluation of Carbothera in the Treatment of Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Mitsubishi-Rayon-Cleansui (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: B2014:037
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2014-09

CONDITIONS: Critical Lower Limb Ischemia; Critical Limb Ischemia; Foot Ulcer; Skin Ulceration
Keywords: Critical Limb Ischemia; Limb Ischemia; Wound Care; Hemodialysis; Dialysis; Skin Ulceration
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Foot Ulcer; Skin Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CO2-Enriched Tap Water (Carbothera) (Experimental): CO2-enriched tap water (CO2 concentration, 1000-1200 ppm) maintained at a temperature of 37˚C. Tap water will be enriched with CO2 by the investigational Carbothera device.
  Interventions: Procedure: CO2-Enriched Tap Water (Carbothera)
- Non-CO2-Enriched Tap Water (Placebo Comparator): Non-CO2-enriched tap water (i.e. normal tap water) maintained at a temperature of 37˚C.
  Interventions: Procedure: Non-CO2-Enriched Tap Water

INTERVENTIONS:
Procedure: CO2-Enriched Tap Water (Carbothera) — Participants will undergo foot bathing with CO2-enriched tap water (CO2 concentration, 1000-1200 ppm) maintained at a temperature of 37˚C with an immersion time of 15 mins, 3 times per week for 4 consecutive months. Participants will be rested on a chair for 15 min before foot bathing. If participant is undergoing hemodialysis, foot bathing will occur prior to their routine hemodialysis procedure.
  Arms: CO2-Enriched Tap Water (Carbothera)
Procedure: Non-CO2-Enriched Tap Water — Participants will undergo foot bathing with non-CO2-enriched tap water maintained at a temperature of 37˚C with an immersion time of 15 mins, 3 times per week for 4 consecutive months. Participants will be rested on a chair for 15 min before foot bathing. If participant is undergoing hemodialysis, foot bathing will occur prior to their routine hemodialysis procedure.
  Arms: Non-CO2-Enriched Tap Water

SUMMARY:
Foot ulceration usually precedes more serious foot complications such as infection, gangrene or amputation. The risk of developing foot ulcers has been estimated to be higher in individuals with kidney disease. Patients with kidney disease receiving dialysis have an increased prevalence of critical limb ischemia. Carbon dioxide (CO2) foot bathing has been reported to improve subcutaneous microcirculation. The proposed clinical study will evaluate the therapeutic potential of CO2 enriched water (produced by the Carbothera device) on treating foot ulcers in patients with critical limb ischemia and undergoing hemodialysis. Forty individuals how have a distal extremity ulcer who are currently undergoing hemodialysis will participate in this study.

DETAILED DESCRIPTION:
This is a multi-centered, placebo controlled and randomized clinical study designed to evaluate the therapeutic potential of CO2 enriched water on the treatment of distal extremity (foot) ulcers in patients with critical limb ischemia undergoing hemodialysis. Study participants will be patients receiving dialysis at two local hospitals in Winnipeg and will have been diagnosed with CLI and foot ulceration. Patients will be randomized to receive either treatment with CO2-enriched tap water, 1,000-1200 ppm CO2 (TREATMENT GROUP), or non-enriched tap water (CONTROL GROUP), bath therapy at 37ºC on the same day as dialysis (typically 3 times/wk), for 15 min for 4 months,. Blood (approximately 20 ml) will also be collected at baseline and at the end of every month of the treatment period (for a total of 5 collections) for the measurement of the different biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants ≥ 18 years of age with at least one distal extremity ulcer (arterial ischemic ulcer).
2. No acute medical illness and on conventional medical management prior to Carbothera.
3. Willingness and ability to provide written informed consent

Exclusion Criteria:

1. DVT or PE within 12 months.
2. Subjects with known active cancer, HIV, hepatitis B virus, hepatitis C virus, human transmissible spongiform encephalopathy, Treponema pallidum.
3. Subjects who are deemed to have an infection of the distal extremity ulcer.
4. Women who are pregnant
5. Unstable angina.
6. Acute MI within 1 month.
7. Stroke within 1 month.
8. Patient scheduled for revascularization during the 4-month intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Ulceration Area, Volume, Depth and Rate | 4 months
  Measurement of ulceration area, volume, depth and rate will be completed at Baseline (Day 1), Week 4, Week 8, Week 12 and Week 16 using an approved (Health Canada) portable hand-held 3D digital wound imaging camera (SilhouetteStar from Aranz Medical, New Zealand).
Changes in Ankle Brachial Index (ABI)/Blood Flow | 4 Months
  A continuous wave, hand held Doppler machine will be used with a blood pressure cuff and a conventional sphygmomanometer to measure the systolic pressure in both the posterior tibial (PT) and dorsalis pedis (DP) arteries. If no PT or DP arterial signals are found, the anterior tibial and/or peroneal artery pressure will be recorded. The ankle systolic pressure and brachial systolic blood pressure will be calculated as ankle systolic pressure/bronchial systolic pressure (ABI). The subject will be asked to rest supine for 10 minutes before ABI measurements. Brachial systolic and diastolic pressures as well as heart rate will be measured. Measurement of ABI will be conducted at Baseline (Day 1), and at weeks 4, 8, 12 and 16.

SECONDARY OUTCOMES:
Changes in Degree of Rest Pain | 4 Months
  Changes in the degree of rest pain will be measured using the McGill Pain Questionnaire which will be administered at Baseline (Day 1), Weeks 8 and 16.
Changes Limb Oxygenation | 4 Months
  Changes in limb blood volume and oxygenation will be recorded using noninvasive near infra-red spectroscopy (NIRS). NIRS measures the percentage of hemoglobin oxygen saturation in the microcirculation of tissue up to 3 cm below the skin.
Changes in Angiogenesis Marker: vascular endothelial growth factor (VEGF) | 4 Months
  A fasting blood sample will be obtained from the participant at the Baseline Visit (Day 1), and Weeks 4, 8, 12 and 16 visits for the purpose of measurement of the angiogenesis marker: vascular endothelial growth factor (VEGF).
Changes in Inflammatory Markers: TNFα, IL-6 and C - reactive protein | 4 Months
  A fasting blood sample will be obtained from the participant at the Baseline Visit (Day 1), and Weeks 4, 8, 12 and 16 visits for the purpose of measurement of inflammatory markers: TNFα, IL-6 and C - reactive protein.
Changes in Markers of Glucose Handling: HbA1c and Fasting Blood Glucose | 4 Months
  A fasting blood sample will be obtained from the participant at the Baseline Visit (Day 1), and Weeks 4, 8, 12 and 16 visits for the purpose of measurement of blood glucose and glycated hemoglobin (hemoglobin A1c).
Changes in Lipid Profile | 4 Months
  A fasting blood sample will be obtained from the participant at the Baseline Visit (Day 1), and Weeks 4, 8, 12 and 16 visits for the purpose of measurement of the participant's lipid profile, specifically, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides.
Changes in Use of Bespoke Footwear and/or ability to Walk Barefoot | 4 Months
  A patient self-report on the use of bespoke footwear or insoles and the ability to walk barefoot at home will be obtained at the Baseline Visit (Day 1) and at Weeks 8 and 16.
Incidence of Amputation | 4 Months
  Incidence of amputation of the distal extremity under study will be monitored during participation in the study.
Use of Antibiotics Indicated for the Ulcer Treatment | 4 Months
  Use of antibiotics indicated for the ulcer treatment during the period of the trial will also be recorded in a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Amarjit S Arneja, MD, Principal Investigator — St. Boniface Hospital
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Sciences Centre- Rehabilitation Hospital, Winnipeg, Manitoba

REFERENCES:
- [Background] Alnaeb ME, Crabtree VP, Boutin A, Mikhailidis DP, Seifalian AM, Hamilton G. Prospective assessment of lower-extremity peripheral arterial disease in diabetic patients using a novel automated optical device. Angiology. 2007 Oct-Nov;58(5):579-85. doi: 10.1177/0003319707305685. PMID 18024941
- [Background] Beckert S, Sundermann K, Wolf S, Konigsrainer A, Coerper S. Haemodialysis is associated with changes in cutaneous microcirculation in diabetes mellitus. Diabet Med. 2009 Jan;26(1):89-92. doi: 10.1111/j.1464-5491.2008.02610.x. PMID 19125767
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] Fellahi JL, Butin G, Zamparini G, Fischer MO, Gerard JL, Hanouz JL. Lower limb peripheral NIRS parameters during a vascular occlusion test: an experimental study in healthy volunteers. Ann Fr Anesth Reanim. 2014 Jan;33(1):e9-14. doi: 10.1016/j.annfar.2013.11.014. Epub 2013 Dec 27. PMID 24373673
- [Background] Game FL, Chipchase SY, Hubbard R, Burden RP, Jeffcoate WJ. Temporal association between the incidence of foot ulceration and the start of dialysis in diabetes mellitus. Nephrol Dial Transplant. 2006 Nov;21(11):3207-10. doi: 10.1093/ndt/gfl427. Epub 2006 Jul 28. PMID 16877485
- [Background] Hartmann BR, Bassenge E, Hartmann M. Effects of serial percutaneous application of carbon dioxide in intermittent claudication: results of a controlled trial. Angiology. 1997 Nov;48(11):957-63. doi: 10.1177/000331979704801104. PMID 9373047
- [Background] Hayashi H, Yamada S, Kumada Y, Matsuo H, Toriyama T, Kawahara H. Immersing Feet in Carbon Dioxide-enriched Water Prevents Expansion and Formation of Ischemic Ulcers after Surgical Revascularization in Diabetic Patients with Critical Limb Ischemia. Ann Vasc Dis. 2008;1(2):111-7. doi: 10.3400/avd.AVDoa08001. Epub 2008 Oct 24. PMID 23555347
- [Background] McGrath NM, Curran BA. Recent commencement of dialysis is a risk factor for lower-extremity amputation in a high-risk diabetic population. Diabetes Care. 2000 Mar;23(3):432-3. doi: 10.2337/diacare.23.3.432. No abstract available. PMID 10868890
- [Background] Ndip A, Rutter MK, Vileikyte L, Vardhan A, Asari A, Jameel M, Tahir HA, Lavery LA, Boulton AJ. Dialysis treatment is an independent risk factor for foot ulceration in patients with diabetes and stage 4 or 5 chronic kidney disease. Diabetes Care. 2010 Aug;33(8):1811-6. doi: 10.2337/dc10-0255. Epub 2010 May 18. PMID 20484126
- [Background] Nishimura N, Sugenoya J, Matsumoto T, Kato M, Sakakibara H, Nishiyama T, Inukai Y, Okagawa T, Ogata A. Effects of repeated carbon dioxide-rich water bathing on core temperature, cutaneous blood flow and thermal sensation. Eur J Appl Physiol. 2002 Aug;87(4-5):337-42. doi: 10.1007/s00421-002-0626-0. Epub 2002 Jun 7. PMID 12172871
- [Background] Rogers LC, Bevilacqua NJ, Armstrong DG, Andros G. Digital planimetry results in more accurate wound measurements: a comparison to standard ruler measurements. J Diabetes Sci Technol. 2010 Jul 1;4(4):799-802. doi: 10.1177/193229681000400405. PMID 20663440
- [Background] Shuler MS, Reisman WM, Whitesides TE Jr, Kinsey TL, Hammerberg EM, Davila MG, Moore TJ. Near-infrared spectroscopy in lower extremity trauma. J Bone Joint Surg Am. 2009 Jun;91(6):1360-8. doi: 10.2106/JBJS.H.00347. PMID 19487513
- [Background] Toriyama T, Kumada Y, Matsubara T, Murata A, Ogino A, Hayashi H, Nakashima H, Takahashi H, Matsuo H, Kawahara H. Effect of artificial carbon dioxide foot bathing on critical limb ischemia (Fontaine IV) in peripheral arterial disease patients. Int Angiol. 2002 Dec;21(4):367-73. PMID 12518118
- [Background] Wakimoto MM, Kadosaki M, Nagata H, Suzuki KS. The usefulness of near-infrared spectroscopy in the anesthetic management of endovascular aortic aneurysm repair. J Anesth. 2012 Dec;26(6):932-5. doi: 10.1007/s00540-012-1435-1. Epub 2012 Jun 26. PMID 22733429
- [Background] Dachun Xu, Jue Li, Liling Zou, Yawei Xu, Dayi Hu, Pagoto SL, Yunsheng Ma. Sensitivity and specificity of the ankle--brachial index to diagnose peripheral artery disease: a structured review. Vasc Med. 2010 Oct;15(5):361-9. doi: 10.1177/1358863X10378376. PMID 20926495
- [Background] Zhang Q, Lindberg LG, Kadefors R, Styf J. A non-invasive measure of changes in blood flow in the human anterior tibial muscle. Eur J Appl Physiol. 2001 May;84(5):448-52. doi: 10.1007/s004210100413. PMID 11417434
- See also: St. Boniface Hospital Research Centre — http://www.sbrc.ca
- See also: St. Boniface Hospital — http://www.sbgh.mb.ca